CLINICAL TRIAL: NCT01493063
Title: BRD/11/02-Y "LACTACOL 01 - Impact of Breast Milk on the Neurodevelopment of Preterm Newborns".
Brief Title: LACTACOL 01 - Impact of Breast Milk on the Neurodevelopment of Preterm Newborns
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/11/02-Y
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Prematurity of Fetus
Keywords: preterm infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breastmilk samples et infant serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physiopathology — Samples of breastmilk and infant serum and questionnaires.

SUMMARY:
The aim of the study is to estimate the impact of the protein content of breastmilk at the end of hospitalization of the preterm newborn, on the neurodevelopment at 2 years old.

The investigators expect a difference of at least 5 points of Development Quotient (DQ) when comparing extreme terciles of the protein content of breastmilk at the end of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Maternal decision of breastfeeding
* Born between 28 and 34 weeks of amenorrhea
* No important congenital pathology except prematurity
* Efficiency of the breastfeeding compatible with the research by the investigator
* Information and authorization of the parents or the parental authority

Exclusion Criteria:

* Maternal decision of not breastfeeding
* Born before 28 weeks of amenorrhoea or after or at 34 weeks of amenorrhoea
* Important congenital pathology
* Efficiency of the breastfeeding incompatible with the research by the investigator
* Opposition from parents or the parental authority to participate to the research study

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm newborn
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of the protein content of human milk on the neuro-motor development of the preterm infant at 2 years of age | At 2 years of age
  ASQ (Ages and Stages Questionnaires) score at 2 years of age. The calculation of the sample size is only based on this endpoint. We wish to highlight a difference of at least 25 points of the ASQ score between both extreme terciles of protein concentration determined in breast milk at the end of hospitalization, when breastfeeding is exclusive (last sample of breastmilk before the end of hospitalization).

SECONDARY OUTCOMES:
To assess the impact of the protein content of human milk on the Body composition (% fat/lean mass) | At 2 years of age and at 7-8 years of age
  Body composition (% fat/lean mass)
To assess the impact of the protein content of human milk on feeding behavior | At 2 years of age and at 7-8 years of age
  Dietary behavior
To assess the impact of the protein content of human milk on growth trajectory and metabolic status of the preterm infant | At 2 years of age and at 7-8 years of age
  Staturo-weight growth rate
To assess the impact of the protein content of human milk on the coginitive intelligence of the preterm infant | At 7-8 years of age
  Standardized and validated test WISC V
To assess the impact of the protein content of human milk on the executive functioning of the preterm infant | At 7-8 years of age
  Standardized and validated test FEE
To assess the impact of the protein content of human milk on the executive dysfunction of the preterm infant | At 7-8 years of age
  Standardized and validated test BRIEF battery
To assess the impact of the protein content of human milk on the child's behaviour in the classroom of the preterm infant | At 7-8 years of age
  Standardized and validated test GSA
To assess the impact of the protein content of human milk on the generalist clinical evaluation of the preterm infant | At 7-8 years of age
  Standardized and validated test BMT-i
To assess the impact of the protein content of human milk on the physical activity of the preterm infant | At 7-8 years of age
  Actimeter (ACTIGRAPH®)
To assess the impact of the protein content of human milk on the physical activity of the preterm infant | At 7-8 years of age
  ESTEBAN questionnaire (Santé Publique France).

OTHER OUTCOMES:
Ancillary study 1.To assess the association between maternal eating habits(food intake during lactation estimated using the Food Frequency Questionnaire from the National French birth cohort ELFE), and the nutritional composition of human milk.
  Association criterion between nutritional composition of human milk assessed by content determination of macro- and micronutrients, and omics approaches (metabolomics,…) and FFQ score
Ancillary study 2.To assess the chemical safety of human milk:identification of nutritional and environmental factors that could explain the presence of chemical contaminants
  Level of chemical contamination of the human milk
Ancillary study N°3. Composition of breast milk and preterm infant's metabolic status and growth trajectory during the first weeks of life. Biomarkers identified in breastmilk and infant serum: lipidome, metabolome, miRNome, amino acids, oligosaccharides
  Correlation obtained between nutritional data from breast milk and identified metabolic markers in children.
Ancillary study N°4. Relationship between breast milk nutritional data and clinical data of mother-child dyads.
  Correlation obtained between the data.
Ancillary study N°5. Correlation between breast milk protein concentration and neurological development at 7-8 years of age. | At 7-8 years of age
  Correlation between breast milk protein concentration and neurological development at 7-8 years of age.
Ancillary study N°6. Equation for estimating fat mass (percentage) in children with the new version of the Biody Xpert device from Aminogram.
  Validation of an equation for estimating fat mass (percentage) in children with the new version of the Biody Xpert device from Aminogram, using a BodPod measurement as reference.
Ancillary study N°7. Equation for estimating lean mass (percentage) in children with the new version of the Biody Xpert device from Aminogram.
  Validation of an equation for estimating lean mass (percentage) in children with the new version of the Biody Xpert device from Aminogram, using a BodPod measurement as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Boscher, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- University Hospital of Nantes, Nantes, France

REFERENCES:
- [Background] Boquien CY, Billard H, Simon L, Boscher C, Legrand A, Joram E, Moyon T, Alexandre-Gouabau MC, Darmaun D, Roze JC. Breast milk protein content at week 3 after birth and neurodevelopmental outcome in preterm infants fed fortified breast milk. Eur J Nutr. 2021 Oct;60(7):3959-3969. doi: 10.1007/s00394-021-02562-8. Epub 2021 Apr 30. PMID 33929587
- [Derived] Alexandre-Gouabau MC, Moyon T, Douarec C, Moulazem Y, Croyal M, Gourdel M, Roze JC, Simon L, Boscher C, Billard H, David-Sochard A, Reze S, Misery B, Bizec BL, Guillou S, Antignac JP, Boquien CY, Vigneau E, Mahieu B, Cano-Sancho G. An Exploration of the Breast Milk Nutriome, Exposome and Microbiome and their Links to Early Growth in Preterm Infants. J Nutr Biochem. 2026 Jan 14:110268. doi: 10.1016/j.jnutbio.2026.110268. Online ahead of print. PMID 41544718